CLINICAL TRIAL: NCT03154905
Title: The Role of Peripheral and Tissue Chitinase 3-like 1 Protein (YKL 40) Levels as a Bio-marker for Gastrointestinal and Liver Disease
Brief Title: The Role of Peripheral and Tissue Chitinase 3-like 1 Protein Levels as a Bio-marker in IBD
Status: Completed | Type: Observational
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Prof. Eran Goldin, Chairman, Digestive Diseases Institute, Shaare Zedek Medical Center
Other Study IDs: 3287-02-01
Record Dates: First submitted 2013-07-02; First posted 2017-05-16 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The study allows the measurements of chitinase 3 like 1 proteins in blood and tissues. Upon consenting to participation in the study, each volunteer may consent to specimens' storage and additional testing. Even though the samples contain DNA, and participation may include analysis in the RNA level, direct DNA sequencing will not be performed and is not included in the additional testing permitted by the subject.

GROUPS / COHORTS (2):
- Control: Healthy controls
- Study group: Patient diagnosed with any disorder of the digestive system (including the alimentary tract, hepatobiliary tree, pancreas, insulin resistance or diabetes, obesity or malnutrition)

SUMMARY:
The digestive system may be involved in various pathologic conditions, with different inflammatory, metaplastic and neoplastic aspects. As the therapeutic tool-box for digestive diseases grows and becomes more focused, at times targeting specific molecules, decision making in managing patients becomes more and more important, and must be evidence based.

Defining biomarkers with predictive value will theoretically allow physicians in making diagnosis, deciding on a suitable first line therapy (with specific endpoints suggesting response or indicating 2nd line therapy is indicated) and finally may suggest surgical intervention is warranted, thus forming an "individually tailored treatment" for each patient. These biomarkers may be located in the peripheral blood, in the gastrointestinal tract in general, or confined to specific intestinal lesions.

Chitinase 3-like 1 protein (YKL-40) is produced by different tissues (e.g. - synovium, smooth muscle, intestinal epithelium). Its specific action is unknown, but several reports have described it in different inflammatory conditions including those involving the gastrointestinal system. Chitinase 3 like-1 protein (YKL-40) has also been studied for its possible role in angio and onco-genesis.

This study aims to evaluate the diagnostic and prognostic value of peripheral and tissue Chitinase 3-like-1 (YKL 40) levels in gastrointestinal and liver diseases.

DETAILED DESCRIPTION:
For periphery tests: 10 ml blood will be collected from all eligible subjects into SST tubes. Then serum will be separated and freeze at -80 degrees until analysis of Chitinase 3 like-1 protein by ELISA.

For tissue tests: biopsies will be taken from colons of eligible participants. One part of these biopsies will be freeze until analysis of Chitinase 3 like-1 protein by ELISA. The other part of the biopsies will be placed in dishes with appropriate media and will be incubated in 37 degrees in order to follow cytokine secretion for 24 h. Media will be collected after 24 h and then freeze until further analysis of Chitinase 3 like-1 protein by ELISA. The investigators will also measure mRNA levels of Chitinase 3 like-1 protein in collected biopsies.

The investigators will try to correlate between the Chitinase 3 like-1 protein levels in the blood and in tissue among various groups of participants and will compare between healthy participants and IBD participants. The investigators will also follow mRNA expression in tissue biopsies taken from all the participants.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Signed informed consent
* Any patient followed or treated by the digestive disease institute team (including ambulatory, hospitalized or undergoing procedure, endoscopy, surgery, endovascular or biopsy).

Exclusion Criteria:

* Pregnancy
* Inability to obtain informed consent
* Bleeding diathesis or any other condition precluding tissue biopsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any patient diagnosed with any disorder of the digestive system (including the alimentary tract, hepatobiliary tree, pancreas, insulin resistance or diabetes, obesity or malnutrition)
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-02; Primary Completion 2014-12 (Actual); Study Completion 2016-01-09 (Actual)

PRIMARY OUTCOMES:
Chitinase 3-like-1 (YKL 40) levels measured by ELISA | 5 years
  ELISA will be used to determine the blood levels and biopsies (organ cultures) levels of Chitinase 3-like-1

CONTACTS AND LOCATIONS:
Overall Officials: Eran Goldin, MD, Principal Investigator — Shaare Zedek Medical Center, Jerusalem, Israel
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No